CLINICAL TRIAL: NCT05200741
Title: A Randomized, Double-blinded, Placebo-controlled Study to Evaluate the Safety and Immunogenicity of DelNS1-2019-nCoV-RBD-OPT1 as Booster Vaccine for COVID-19 in Healthy Adults Who Have Received 2 Doses of BNT162b2
Brief Title: To Evaluate Safety & Immunogenicity of DelNS1-2019-nCoV-RBD-OPT1 for COVID-19 in Healthy Adults Received 2 Doses of BNT162b2
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CTC2235
Record Dates: First submitted 2022-01-20; First posted 2022-01-21 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-01

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Product (Experimental): DelNS1-2019-nCoV-RBD-OPT1 virus titre at not less than 6.3 lg CCID50/dose, 2 doses 3 weeks apart, intranasal administration
  Interventions: Biological: DelNS1-2019-nCoV-RBD-OPT1
- Reference Product (Placebo Comparator): Matching placebo, 2 doses 3 weeks apart, intranasal administration
  Interventions: Biological: Matching placebo

INTERVENTIONS:
Biological: DelNS1-2019-nCoV-RBD-OPT1 — Influenza Virus Vector COVID-19 Vaccine for Intranasal Spray
  Arms: Test Product
Biological: Matching placebo — Solution for Intranasal Spray
  Arms: Reference Product

SUMMARY:
To evaluate the safety and immunogenicity of DelNS1-2019-nCoV-RBD-OPT1 as booster vaccine for COVID-19 in healthy adults who have received 2 doses of BNT162b2

DETAILED DESCRIPTION:
This is a randomized, double-blinded, placebo-controlled study to evaluate the safety and immunogenicity of DelNS1-2019-nCoV-RBD-OPT1 as booster vaccine for COVID-19 in healthy adults who have received 2 doses of BNT162b2. Each subject will receive 2 vaccinations or matching placebo 3 weeks apart.

ELIGIBILITY:
Inclusion Criteria:

1. Informed Consent: The subject (or the subject's legally acceptable representative, if applicable) must be capable of giving written informed consent and, prior to the commencement of any study-specific procedure, must sign an ICF indicating the consent on the subject's voluntary participation in the study and compliance with the requirements and restrictions listed on the ICF.
2. BNT162b2 Vaccination Status: The subject must have received 2 doses of BNT162b2 in Hong Kong, with the second dose completed at least 180 days prior to the first vaccination.
3. Gender and Age: Male or female, at the age of ≥ 18 and ≤ 75 on the day of signing the ICF.
4. Body Weight and BMI: Body weight ≥ 45 kg and BMI ≥ 18.5 kg/m2 and < 25 kg/m2 at screening and baseline.
5. Medical Conditions or Diagnoses: Existence of all of the following medical conditions or diagnoses:

   1. Generally in good health with no clinically significant abnormality, as determined by medical history, physical examination, 12-lead ECG and clinical laboratory tests at screening and baseline;
   2. Normal vital signs at screening and baseline, as defined by:

      * Body (tympanic) temperature ≤ 37.5 oC;
      * Resting pulse rate ≥ 50 and ≤ 100 bpm; and
      * DBP ≥ 50 and ≤ 90 mmHg and SBP ≥ 90 and ≤ 140 mmHg.
6. Contraception: Willingness and agreement to undertake measures to avoid pregnancy of the subject or the subject's sexual partner(s) as detailed below:

   1. A female subject who is a woman of childbearing potential (WOCBP) must be willing and agree to remain abstinent or practise at least one effective contraceptive method from at least 30 days prior to the first vaccination until 60 days after the second vaccination;
   2. A male subject (i) who is sexually active with a WOCBP (except who is permanently sterile by bilateral orchiectomy or vasectomy) must be willing and agree to remain abstinent or practise at least one effective contraceptive method from the first vaccination until 60 days after the second vaccination; and (ii) must be willing and agree to refrain from sperm donation during the aforesaid period.
7. Breastfeeding: A female subject must be willing and agree to avoid engagement in breastfeeding at any time from the first vaccination until 60 days after the second vaccination.
8. Blood Donation: Willingness and agreement to avoid blood donation from screening to the end of the period of participation in this study.

Exclusion Criteria:

1. Medical History: History of any of the following diseases or conditions:

   1. COVID-19;
   2. SARS;
   3. Any significant respiratory diseases (e.g. COPD, asthma);
   4. Any significant cardiovascular disease (e.g. angina, cardiac arrhythmias);
   5. Blood dyscrasias or any significant disorder of coagulation;
   6. Any chronic liver disease (e.g. autoimmune hepatitis and cirrhosis);
   7. Any chronic infection (e.g. hepatitis B, hepatitis C and HIV);
   8. Any malignant neoplastic disease;
   9. Encephalopathy, neuropathy or unstable central nervous system (CNS) pathology;
   10. Any psychiatric disorder, psychotic disorder, major affective disorder or suicidal ideation;
   11. Any immunodeficiency or autoimmune disease;
   12. Any severe allergic reaction (e.g. anaphylaxis) to any vaccine or substance, which requires hospitalization or emergency medical care;
   13. Any nasal septal defect, cleft palate, nasal polyps or other nasal abnormality that might affect vaccine administration;
   14. History of alcohol or illicit drug abuse, or used any illicit drug within 6 months prior to screening.
2. Medical Conditions or Diagnoses: Existence of any of the following medical conditions or diagnoses:

   1. Positive serum pregnancy test at screening or positive urine pregnancy test at baseline (for WOCBP);
   2. IgE level > 1,000 IU/ml at screening;
   3. Positive SARS-CoV-2 test result in deep throat saliva (DTS) within 4 days prior to the first vaccination;
   4. Positive HIV test result at screening;
   5. Positive HBsAg test result at screening;
   6. Positive HCV antibody test result at screening;
   7. Positive urine drug screen test result or positive blood alcohol test result at screening or baseline;
   8. Clinically significant abnormality of T3, T4 or TSH at screening;
   9. Clinically significant abnormality of PT (INR) or aPTT at screening.
3. Prior/Concomitant Interventions: Use of or undergoing any of the following prior or concomitant medications, therapies or interventions:

   1. Any COVID-19 or coronavirus vaccine at any time prior to the first vaccination, except BNT162b2 or planned use of any such vaccine throughout the study;
   2. Any vaccine other than COVID-19 or coronavirus vaccines within 28 days prior to the first vaccination, or planned use of any such vaccine up to 28 days after the second vaccination;
   3. Any immune-modifying medication/therapy (e.g. immunomodulator and immunosuppressant) within 6 months prior to the first vaccination, or planned use of any such medication/therapy throughout the study;
   4. Any blood product (including blood transfusion) or immunoglobulin within 3 months prior to the first vaccination, or planned use of any such therapy throughout the study;
   5. Any anticoagulation medication within 28 days prior to the first vaccination, or planned use of any such medication up to 28 days after the second vaccination;
   6. Any psychotropic medication within 28 days prior to the first vaccination, or planned use of any such medication up to 28 days after the second vaccination;
   7. Regular use of any inhaled/nebulized corticosteroid;
   8. Any intranasal preparation within 48 hours prior to the first vaccination, or planned use of any such preparation up to 48 hours after the second vaccination;
   9. Any influenza antiviral medication within 48 hours prior to the first vaccination, or planned use of any such medication up to 14 days after the second vaccination;
   10. Any prescription or over-the-counter medication within 7 days prior to the first vaccination, unless with the investigator's approval;
   11. Donated ≥ 450 ml of blood within 28 days prior to the first vaccination;
   12. Prior nasal surgery or nasal cauterization.
4. Prior/Concurrent Clinical Study: Prior or concurrent participation in any other clinical study, including:

   1. Prior or current participation in another COVID-19 vaccine study;
   2. Prior participation in any interventional clinical study and use of any investigational intervention within 90 days prior to the first vaccination;
   3. Concurrent participation or plan for participation in another interventional clinical study during participation in this study.
5. Other Significant Medical Conditions: Any clinically significant concomitant disease or condition that, in the reasonable opinion of the investigator, may interfere with the subject's participation in this study or pose an unacceptable safety risk for the subject's participation in this study.
6. Special Conditions: Existence of any of the following special conditions:

   1. Close contact with anyone known to have COVID-19 within 30 days prior to the first vaccination;
   2. Travelled outside Hong Kong within 14 days prior to the first vaccination;
   3. Planned to travel outside Hong Kong at any time during the period from screening to Day 50(±3) visit.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-02-08 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Reactogenicity | Day 1 to 15 and Day 22 to 36
  Occurrence of solicited local events (nasal irritation, sneezing, nasal congestion, cough, sore throat, change in smell, change in taste, change in vision and eye pain) and solicited systemic events (fever, headache, malaise, myalgia, joint pain, nausea, vomiting, diarrhea, abdominal pain, chills and sweating) for a 14-day period after each vaccination
Adverse Events | Day 1 to Day 202(±7)
  Occurrence of unsolicited AEs, Serious Adverse Events (SAEs) and Adverse Events of Special Interest (AESIs)
Neutralizing Antibodies in Serum against Live SARS-CoV-2 Measured by Neutralization Assay | Day 1(pre-dose), 22(pre-dose), 36(+2) and 50(±3)
  Measurement of neutralizing antibody levels by microneutralization (MN) assay in serum samples
Binding Antibodies in Serum against SARS-CoV-2 RBD Measured by CMIA | Day 1(pre-dose), 22(pre-dose), 36(+2) and 50(±3)
  Measurement of binding antibody responses by chemiluminescent microparticle immunoassay (CMIA) in serum samples

SECONDARY OUTCOMES:
T-cell Responses against SARS-CoV-2 Spike Peptide Measured by ELISpot | Day 1(pre-dose), 22(pre-dose), 36(+2) and 50(±3)
  Enumeration of antigen-specific T cells by IFN gamma ELISpot assay in serum samples
Total Ig Antibodies in Mucosal Secretion against SARS-CoV-2 RBD Measured by ELISA | Day 1(pre-dose), 4(+1), 22(pre-dose), 25(+1), 36(+2) and 50(±3)
  Measurement of total Ig antibody levels in saliva samples

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Fan-ngai Hung, Principal Investigator — The University of Hong Kong
Locations (1):
- HKU Phase 1 Clinical Trials Centre, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
The results of this study will be publicly disseminated by ways of publication(s) in peer-reviewed scientific journal(s), presentation(s) in scientific conference(s), posting on public clinical trial registry(ies) and/or otherwise instead of individual participant data (IPD) sharing.

REFERENCES:
- [Background] Influenza Virus Vector COVID-19 Vaccine for Intranasal Spray (DelNS1-2019-nCoV-RBD-OPT1) Phase III Clinical Trial - Investigator's Brochure (Version 2.0, Dated 02-Sep-2021).
- [Background] Wang P, Zheng M, Lau SY, Chen P, Mok BW, Liu S, Liu H, Huang X, Cremin CJ, Song W, Chen Y, Wong YC, Huang H, To KK, Chen Z, Xia N, Yuen KY, Chen H. Generation of DelNS1 Influenza Viruses: a Strategy for Optimizing Live Attenuated Influenza Vaccines. mBio. 2019 Sep 17;10(5):e02180-19. doi: 10.1128/mBio.02180-19. PMID 31530680
- [Background] Zheng M, Wang P, Song W, Lau SY, Liu S, Huang X, Mok BW, Liu YC, Chen Y, Yuen KY, Chen H. An A14U Substitution in the 3' Noncoding Region of the M Segment of Viral RNA Supports Replication of Influenza Virus with an NS1 Deletion by Modulating Alternative Splicing of M Segment mRNAs. J Virol. 2015 Oct;89(20):10273-85. doi: 10.1128/JVI.00919-15. Epub 2015 Jul 29. PMID 26223635
- See also: Accessed on 15 November 2021 — https://www.fda.gov/media/139638/download
- See also: Accessed on 15 November 2021 — https://www.fda.gov/downloads/BiologicsBloodVaccines/GuidanceComplianceRegulatoryInformation/Guidances/Vaccines/ucm091977.pdf
- See also: Accessed on 07 January 2021 — https://www.gmp-compliance.org/files/guidemgr/E9-R1_Step4_Guideline_2019_1203.pdf
- See also: Accessed on 15 November 2021 — https://covid19.who.int/table